CLINICAL TRIAL: NCT00570297
Title: Genetic Influences of Albuterol Response In Children With Bronchiolitis
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: UConn Health (Other)
Responsible Party: Sponsor
Other Study IDs: 07-158; UCHC GCRC# 667 (Other: University of Connecticut Health Center)
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2022-10

CONDITIONS: Bronchiolitis
Keywords: Pediatric; Polymorphism, Genetic; Adrenergic beta-Agonists
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bronchiolitis is a significant cause of morbidity and hospitalization in children, accounting for approximately 125,000 hospitalizations per year in the U.S. Recently, genetic variations of the β2-adrenergic receptor (β2-AR) have been shown to influence response to β2-AR agonist therapy in children with asthma. We suspect that genetic variations of the β2-AR also affect response to β2-AR agonist therapy in children with bronchiolitis.

DETAILED DESCRIPTION:
Bronchiolitis is a significant cause of morbidity and hospitalization in children, accounting for approximately 125,000 hospitalizations per year in the U.S. Of these hospitalized children, 8% will require intensive care unit (ICU) admission and 67% of these children will require mechanical ventilation. Mortality in previously healthy children is generally low, however, in children with high-risk medical conditions such as prematurity or congenital heart disease, mortality can be as high as 3%. In addition, bronchiolitis infections are associated with long term respiratory problems including development of recurrent wheezing, airway hyperreactivity, and asthma.

Treatment for bronchiolitis is largely supportive. Despite four decades of clinical trials, there are no therapies demonstrated to be effective in shortening either hospitalization or ICU length of stay in children with bronchiolitis. The use of β2-adrenergic receptor (β2-AR) agonists has received the most attention from investigators, however the results of clinical trials have been contradictory and inconclusive.

Recently, investigators have shown that genetic factors have important influences on a patient's response to β2-AR agonists. Single nucleotide polymorphisms (SNP) at amino acid position 16 of the β2-AR gene are thought to be the most functionally relevant. A change at base 46 from adenine to guanine results in the amino acid sequence of the β2-AR containing a glycine (Gly), rather than an arginine (Arg), at amino acid position 16. Patients homozygous for Gly at this position (Gly/Gly) have been shown to have improved response to β2-AR agonist therapy when compared to children homozygous for Arginine (Arg/Arg) or heterozygous (Arg/Gly). The next most common polymorphism of the β2-AR gene, glutamine to glutamic acid at position 27 (Glu27Gln), may be associated with the development of asthma and airway hyperresponsiveness, but these relationships are less clear.

We believe that genetic factors also influence response to β2-AR agonist therapy in children with bronchiolitis. Specifically, we believe that β2-AR polymorphisms at amino acid position 16 affect response to acute β2-AR agonist therapy in children with bronchiolitis. Our hypothesis is that children with bronchiolitis who are homozygous for glycine at amino acid position 16 (Gly/Gly) will have improved response to inhaled β2-AR agonist therapy.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the CCMC with a primary admission diagnosis of bronchiolitis.
* Age between 0 and 2 years.
* Intubated with cuffed endotracheal tube and mechanically ventilated for less than 72 hours.
* Receiving inhaled albuterol therapy

Exclusion Criteria:

* Congenital Heart Defect
* Immunodeficiency
* Pre-existing chronic lung disease, including asthma
* Receiving additional bronchodilator therapy (such as theophylline or ipratropium) or any therapy that would interfere with measuring pulmonary compliance or resistance
* Receiving Albuterol more frequently than every 4 hours

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children hospitalized in the intensive care unit with bronchiolitis
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2007-12; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in lung resistance | Immediate
  The primary end point is change in lung resistance following a single dose of inhaled b2-AR agonist therapy (albuterol).

SECONDARY OUTCOMES:
Change in lung compliance | Duration of hospitalization
  To assess the change in lung compliance following a single dose of inhaled b2-AR agonist therapy (albuterol)
Comparison by genotype | Duration of Hospitalization
  To compare duration of mechanical ventilation and ICU hospital length of stay by genotype

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Carroll, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No